CLINICAL TRIAL: NCT06775925
Title: Robot-assisted Vs. Conventional Occupational Therapy of the Upper Limb in Individuals with Cervical Spinal Cord Injury: the Armeo X-over Trial
Brief Title: Robot-assisted Vs. Conventional Occupational Therapy of the Upper Limb in Individuals with Cervical Spinal Cord Injury
Acronym: Armeo X-over
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Swiss Paraplegic Research, Nottwil (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 2020-22
Record Dates: First submitted 2024-12-24; First posted 2025-01-15 (Actual); Last update posted 2025-03-10 (Actual); Status verified 2025-03

CONDITIONS: Cervical Spinal Cord Injury
Keywords: upper limb function; robot-assisted therapy; occupational therapy

STUDY DESIGN:
Intervention Model Description: Randomized, assessor-blind, two-period, crossover trial
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- RT-OT (Experimental): A stratified randomisation procedure will be used to allocate the sequence with either RT followed by OT or vice versa. The participants will performe unilateral robot-asssited therapy for 3 x 30 minutes per week for 6 weeks first, and then the unilateral conventional occupational therapy also for 3 x 30 minutes per week for 6 weeks.
  Interventions: Other: Unilateral robot-assisted therapy (RT); Other: Unilateral conventional occupational therapy (OT)
- OT-RT (Experimental): A stratified randomisation procedure will be used to allocate the sequence with either OT followed by RT or vice versa. The participants will perform unilateral conventional occupational therapy for 3 x 30 minutes per week for 6 weeks first, and then unilateral robot-assisted therapy also for 3 x 30 minutes per week for 6 weeks.
  Interventions: Other: Unilateral robot-assisted therapy (RT); Other: Unilateral conventional occupational therapy (OT)

INTERVENTIONS:
Other: Unilateral robot-assisted therapy (RT) — RT will be performed as an add-on therapy to the clinical routine therapy scheme for 3 x 30 minutes per week for 6 weeks. RT is applied using the ArmeoSpring, an exoskeleton that provides adjustable antigravity weight support for the arm through a system of springs (no actuators).
Other: Unilateral conventional occupational therapy (OT) — The OT is applied as add-on therapy for 3 x 30 minutes per week for 6 weeks. OT comprises strengthening exercises (concentric and eccentric) with and without resistance, grasping exercises, fine motor training, peg games, and activity-based tasks which are unilaterally doable.

SUMMARY:
The goal of this clinical trial is to learn the effects of robot-assisted therapy using the ArmeoSpring on upper limb function compared to conventional occupational therpay in individuals with cervical spinal cord injury (cSCI). The main questions it aims to answer are:

- Which of the two forms of therapy, robot-assisted therapy or conventional occupational therapy, is more effective in terms of improving arm and hand function?

The study is designed as a cross-over trial, which means that each participant will receive both therapy forms consecutively, whereas the order is assigned randomly (either robot-assisted therapy first and then occupational therapy, or vice versa).

In addition to their clinical routine therapy , participants will:

* complete a baseline assessment
* practice one therapy form (either robot-assisted or occupational therapy) with one arm for 6 weeks (3 x 30 min per week)
* complete a intermediate assessment
* practice the other therapy form (either occupational or robot-assisted therapy) with one arm for 6 weeks (3 x 30 min per week)
* complete a post assessment
* complete a follow-up assessment (if the post assessment was completed prior to 150 days post-injury)

DETAILED DESCRIPTION:
After cervical spinal cord injury (cSCI), motor and sensory impairments cause limitations in upper limb function which affect performance of activities of daily living (ADLs), independence and, ultimately, restrict participation and quality of life. Previous studies have shown that individuals with tetraplegia consider improvements in upper limb function to be one of the most significant factors in improving their quality of life. Small improvements in upper extremity function through rehabilitation can lead to substantial increases in independence with ADLs, quality of life and community integration. Repetitive and activity-based exercise can facilitate recovery after SCI by inducing practice-dependent brain and spinal plasticity. To achieve high numbers of repetitions, specialised rehabilitation centres apply innovative therapy methods like robot-assisted therapy (RT) aiming to improve upper limb function. Integrating robotic devices into daily clinical practice may save personnel resources while enabling high-intensive and individualised therapy using motivating feedback (e.g., gamification) and allowing for close monitoring of therapy sessions. Evidence suggests that robot-assisted interventions are safe, feasible and can reduce active assistance provided by therapists.

However, the clinical effectiveness of robot-assisted interventions for patients after cSCI has not been proven so far. For the devices used at the Swiss Paraplegic Centre (SPC) for upper extremity therapy after cSCI, there are only two studies to date that have followed a randomised controlled trial (RCT) design, and both were conducted with inadequate methodological quality (e.g. recruitment period one or two years post-injury respectively). This introduces a lot of variance and it thus remains open whether RT and conventional occupational therapy (OT) just have similar effects, or whether potential effects have been blurred due to imprecise study designs. Moreover, while both RCTs used the actively supporting ArmeoPower, internal analyses have shown that the passively supporting ArmeoSpring is the by far mostly used robotic device for training of the upper extremity inhouse. The ArmeoSpring is an instrumented arm orthosis with a spring mechanism (no actuators) for adjustable antigravity weight support for the arm in a large 3D workspace. However, neither of these robotic devices has ever been properly evaluated for clinical effectiveness .

Therefore, the aim of this study is to systematically investigate the effects of robot-assisted therapy (using the ArmeoSpring) on upper limb function compared to conventional occupational therapy in individuals with intermediate (between 2 weeks and 6 months after injury) cSCI.

ELIGIBILITY:
Inclusion Criteria:

* Informed Consent signed by the subject
* Intermediate (>16 days and ≤81 days post-injury) traumatic or non-traumatic cSCI during primary rehabilitation at the Swiss Paraplegic Centre (SPC)
* Neurological level of injury: C1-T1
* American Spinal Injury Association Impairment Scale (AIS): A-D
* Impairment of upper limb function (GRASSP-QtG score unilateral < 25 at baseline t0)
* Ability to sit for 60 minutes and perform training with ArmeoSpring
* Stratification parameters available

Exclusion Criteria:

* Inability to follow the procedures of the investigation
* Severe concomitant neurological disease
* Concomitant neurodegenerative or progressive diseases
* Impairment of upper limb function due to peripheral nerve lesions
* Severe concurrent medical disease or any other issue that in the opinion of the investigator would confound the results
* Orthopedic limitations of the upper limb
* Device specific contraindications
* Participation in other interventional trials

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-02-01 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Grasp performance | Baseline Assessment (week 1), Intermediate Assessment (week 7), Post Assessment (week 14), Follow-up Assessment (week 18)
  Quantitative subtest of Graded Redefined Assessment of Strength, Sensibility, and Prehension (GRASSP-QtG).
  6 GRASSP-QtG tasks in total, each task is graded from 0 (the task cannot be conducted at all) to 5 (the task is conducted without difficulties using the expected grasping pattern and upper limb function is unaffected).

SECONDARY OUTCOMES:
Qualitative upper limb function | Baseline Assessment (week 1), Intermediate Assessment (week 7), Post Assessment (week 14), Follow-up Assessment (week 18)
  Qualitative, sensation and strength subtest of GRASSP. 3 prehension ability tasks, of which each task is graded from 0 (the task cannot be conducted at all) to 4 (the task is conducted without difficulties and appropriate force) for each arm.
Independence in ADL | Baseline Assessment (week 1), Intermediate Assessment (week 7), Post Assessment (week 14), Follow-up Assessment (week 18)
  Spinal Cord Independence Measure III - Self-report (SCIM-SR). The SCIM-SR is assessed in 3 domains. The first domain "Self-Care" consists of 6 items and the scores range from 0 (e.g. full support needed) to 20 (e.g. completely independent). The second domain "Respiration and sphincter management" include 4 items whereas the third domain " Mobility" contain 9 items, both with scores from 0 - 40. Thus, the total score of SCIM-SR ranges from 0 to 100.
Upper Extremity Motor Score | Baseline Assessment (week 1), Intermediate Assessment (week 7), Post Assessment (week 14), Follow-up Assessment (week 18)
  International Standards for the Neurological Classification of Spinal Cord Injury examination (ISNCSCI-UEMS).
  Manual muscle testing of 5 upper extremity movements is conducted and scored. Each score is graded between 0 (no palpable or visible muscle contraction) to 5 (Full range of motion against maximum resistance) by the medical research council scale.
Handgrip strength | Baseline Assessment (week 1), Intermediate Assessment (week 7), Post Assessment (week 14), Follow-up Assessment (week 18)
  dynamometer
Arm control | Baseline Assessment (week 1), Intermediate Assessment (week 7), Post Assessment (week 14), Follow-up Assessment (week 18)
  Instrumented Action Research Arm Test (iARAT)
Therapy intensity | 18 times during the 12 weeks interventions
  amount of movement quantified by inertial measurement units (IMUs)
Intrinsic Motivation | 6 times during the 12 weeks interventions
  Intrinsic Motivation Inventory (IMI). The full IMI includes 45 items distributed across seven subscales, of which the applicable items and subscales can be chosen. Each item is graded between 1 (not at all true) to 7 (very true).

CONTACTS AND LOCATIONS:
Locations (1):
- Swiss Paraplegic Centre, Nottwil, Canton of Lucerne, Switzerland

IPD SHARING:
Plan to Share IPD: Yes
All IPD that underlie results in a publication.
Supporting Information: Study Protocol

REFERENCES:
- [Background] Yozbatiran N, Francisco GE. Robot-assisted Therapy for the Upper Limb after Cervical Spinal Cord Injury. Phys Med Rehabil Clin N Am. 2019 May;30(2):367-384. doi: 10.1016/j.pmr.2018.12.008. Epub 2019 Mar 2. PMID 30954153
- [Background] Snoek GJ, IJzerman MJ, Hermens HJ, Maxwell D, Biering-Sorensen F. Survey of the needs of patients with spinal cord injury: impact and priority for improvement in hand function in tetraplegics. Spinal Cord. 2004 Sep;42(9):526-32. doi: 10.1038/sj.sc.3101638. PMID 15224087
- [Background] Singh H, Unger J, Zariffa J, Pakosh M, Jaglal S, Craven BC, Musselman KE. Robot-assisted upper extremity rehabilitation for cervical spinal cord injuries: a systematic scoping review. Disabil Rehabil Assist Technol. 2018 Oct;13(7):704-715. doi: 10.1080/17483107.2018.1425747. Epub 2018 Jan 15. PMID 29334467
- [Background] Lynskey JV, Belanger A, Jung R. Activity-dependent plasticity in spinal cord injury. J Rehabil Res Dev. 2008;45(2):229-40. doi: 10.1682/jrrd.2007.03.0047. PMID 18566941
- [Background] Kuchen DB, Hubacher B, Ladner A, Velstra IM, Widmer M. Technology-Assisted Upper Limb Therapy (TAULT): Evaluation of Clinical Practice at a Specialised Centre for Spinal Cord Injury in Switzerland. Healthcare (Basel). 2023 Nov 28;11(23):3055. doi: 10.3390/healthcare11233055. PMID 38063623
- [Background] Kim J, Lee BS, Lee HJ, Kim HR, Cho DY, Lim JE, Kim JJ, Kim HY, Han ZA. Clinical efficacy of upper limb robotic therapy in people with tetraplegia: a pilot randomized controlled trial. Spinal Cord. 2019 Jan;57(1):49-57. doi: 10.1038/s41393-018-0190-z. Epub 2018 Sep 11. PMID 30206423
- [Background] Jung JH, Lee HJ, Cho DY, Lim JE, Lee BS, Kwon SH, Kim HY, Lee SJ. Effects of Combined Upper Limb Robotic Therapy in Patients With Tetraplegic Spinal Cord Injury. Ann Rehabil Med. 2019 Aug;43(4):445-457. doi: 10.5535/arm.2019.43.4.445. Epub 2019 Aug 31. PMID 31499598
- [Background] Anderson KD. Targeting recovery: priorities of the spinal cord-injured population. J Neurotrauma. 2004 Oct;21(10):1371-83. doi: 10.1089/neu.2004.21.1371. PMID 15672628